CLINICAL TRIAL: NCT04105621
Title: Westlake Personalized Nutrition and Health Cohort for Drug Addicts
Acronym: WePN-DA
Status: Completed | Type: Observational
Sponsor: Westlake University (Other)
Collaborators: Zhejiang Drug Rehabilitation Administration (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20190812ZJS0009
Record Dates: First submitted 2019-09-01; First posted 2019-09-26 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-10

CONDITIONS: Drug Addiction; Undernutrition; Drug Abuse
Keywords: Personalized nutrition; Drug addicts; Gut microbiota
MeSH Terms: conditions — Substance-Related Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting venous blood, urine, saliva and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug addicts: This group included drug addicts lived in drug rehablitation center.
- Healthy population: We recruited the healthy participants from the Westlake N-of-1 Trials for Macronutrient Intake (NCT04125602) as healthy control

SUMMARY:
This is a prospective cohort study of drug addicts confined in Zhejiang rehabilitation centers. The primary aim of this study is to investigate the association between diet and health status among drug addicts. The second aim is to characterize the continuous blood glucose response to dietary intakes over 2 weeks. The third aim is to describe the dynamic changes of gut microbiota at three time points in drug addicts during compulsory detoxification and to evaluate the association between gut microbiota, diet and addiction severity.

DETAILED DESCRIPTION:
Over recent decades, there is a growing trend of drug addiction in China that poses great public health challenges. Drug abuse can lead to many health related problems such as malnutrition and mental disorders along with reduced quality of life. Dietary intervention plays a pivotal role in disease prevention and drug rehabilitation for drug addicts, but the associations between dietary intake and health related outcomes among drug addicts remain unclear.

In addition, the relationship between the human gut microbiota and its response to addictive drugs as a newly arisen subject is given wide attention in recent years. However, the underlying mechanism requires further investigation. The dynamic changes of gut microbiota among drug addicts during compulsory drug rehabilitation period are in vague.

Under the same diet exposure, different drug addicts may have different blood glucose responses as well as gut microbiota profiles. Therefore, in order to examine the association between diet, gut microbiota and drug addiction, our study design will include three components: (1) the measurement of dietary intake using FFQ while the menu offered by drug rehabilitation center and food diary; (2) the measurements of blood glucose over 2 weeks using continuous glucose monitors; and (3) the measurements of gut microbiota at three time points using 16s rRNA sequencing techniques.

ELIGIBILITY:
Inclusion Criteria:

* Drug addicts aged between 18 yrs and 65yrs.
* Drug addicts lived in Zhejiang drug rehabilitation centers.
* Drug addicts who have stayed in drug rehabilitation center for no more than 6 months.

Exclusion Criteria:

* Drug addicts diagnosed with cancer or other serious physical and mental disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Drug addicts confined in Zhejiang drug rehabilitation centers will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Continuous blood glucose profile over 2 weeks | Two weeks after enrollment
  Glucose levels were measured using continuous glucose monitoring over 2 week
The dynamic change of gut microbiota within one year | One year after enrollment; includes three sampling time points: baseline, 6 months after enrollment and 12 months after enrollment.
  Fecal microbiota was analyzed using16S rRNA gene sequencing technique

SECONDARY OUTCOMES:
Drug craving intensity | Baseline; 6 months after enrollment; 12 months after enrollment
  This was evaluated by Obsessive Compulsive Drug Use Scale (OCDUS). This scale had 13 items, each with a 5-point Likert-response (1, 2, 3, 4 and 5). Items 6 and 13 were reverse-scored. The total score ranges from 13 to 65 and a higher value represent a higher intensity of drug craving.
The change of BMI | Baseline; 6 months after enrollment; 12 months after enrollment
  BMI in kg/m^2
Nutritional status | Baseline; 6 months after enrollment; 12 months after enrollment
  Nutritional status was measured by mini nutritional assessment (MNA) screening test.
The degree of depression | Baseline; 6 months after enrollment; 12 months after enrollment
  This was evaluated by Beck Depression Inventory-II (BDI-II). Scores in every item of the BDI-II were between 0 and 3. The total score ranges from 0 to 63.
The degree of anxiety | Baseline; 6 months after enrollment; 12 months after enrollment
  This was evaluated by Hamilton Anxiety Scale (HAMA). Scores in every item of the HAMA were between 0 and 4. The total score ranges from 0 to 56.
Body composition | Baseline; 6 months after enrollment; 12 months after enrollment
  Body composition (fat mass, lean mass in kg ) are assessed by bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Zhejiang Drug Rehabilitation Administration, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided